CLINICAL TRIAL: NCT03281226
Title: An Open Label Randomized Phase 2 Clinical Trial to Assess Safety and Tolerability of RIPE vs RIPE Plus N-acetylcysteine in Patients With HIV/Aids and Pulmonary Tuberculosis
Brief Title: RIPE vs RIPE Plus N-acetylcysteine in Patients With HIV/TB Co-infection
Acronym: RIPENACTB
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundação de Medicina Tropical Dr. Heitor Vieira Dourado (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAAE: 60219916.5.0000.0005
Record Dates: First submitted 2017-09-11; First posted 2017-09-13 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Tuberculosis, Pulmonary; HIV/AIDS
Keywords: Pulmonary tuberculosis; HIV/AIDS; Glutathione; N-acetylcysteine; Oxidative stress
MeSH Terms: conditions — Tuberculosis, Pulmonary; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIPE (2m) and RI (4m) (Active Comparator): The patients enrolled in this arm will receive a treatment regimen with an intensive phase lasting two months of rifampicin 150mg + isoniazid 75mg + pyrazinamide 400mg + ethambutol 275mg (combined fixed dose tablet according to the weight) and a continuation with rifampicin 150mg and isoniazid 75mg (combined fixed dose tablet according to the weight) for 4 months.
  Interventions: Drug: RIPE (2m) and RI (4m)
- RIPE+NAC (2m) and RI (4m) (Experimental): The patients enrolled in this arm will receive a treatment regimen with an intensive phase lasting two months of rifampicin 150 mg + isoniazid 75 mg + pyrazinamide 400 mg + ethambutol 275mg (combined fixed dose tablet according to the weight) plus N-acetylcysteine (NAC) and a continuation with rifampicin 150mg and isoniazid 75mg (combined fixed dose tablet according to the weight) for 4 months. The NAC is administered by means of effervescent tablet 1200 mg (two sachets of 600 mg) to be diluted in 200ml of water and administered in a 12-hour interval.
  Interventions: Drug: RIPE+NAC (2m) and RI (4m)

INTERVENTIONS:
Drug: RIPE (2m) and RI (4m) — Rifampicin 150mg + isoniazid 75mg + pyrazinamide 400mg + ethambutol 275mg (oral combined fixed dose tablet according to the weight) for 2 months and a continuation with rifampicin 150mg and isoniazid 75mg (oral combined fixed dose tablet according to the weight) for 4 months
  Arms: RIPE (2m) and RI (4m)
Drug: RIPE+NAC (2m) and RI (4m) — Rifampicin 150 mg + isoniazid 75 mg + pyrazinamide 400 mg + ethambutol 275mg (oral combined fixed dose tablet according to the weight) plus oral N-acetylcysteine (NAC) 1200 mg (600mg twice daily) for 2 months and a continuation with rifampicin 150mg and isoniazid 75mg (oral combined fixed dose tablet according to the weight) for 4 months
  Arms: RIPE+NAC (2m) and RI (4m)

SUMMARY:
Although tuberculosis is a treatable disease, it is currently the infectious disease with the highest mortality in the world. It is estimated that one-third of the world's population is infected. HIV is the main predisposing factor for TB development. The Brazilian Ministry of Health and the World Health Organization recommends that patients should initially be treated orally with RIPE - rifampicin (R), isoniazid (I), pyrazinamide (P) and ethambutol (E). The N-acetylcysteine (NAC) first benefit was reported during the 1960s, when it proved to be an effective mucolytic agent in individuals with cystic fibrosis. Later, a new role arose when investigating its therapeutic potential in acetaminophen intoxication. Cleavage of the acetyl group makes cysteine available for later incorporation into glutathione synthesis, decreased in hepatic injury caused by acetaminophen. This mechanism causes NAC to have an indirect antioxidant effect, which aroused an interest in studying the effect in diseases that occur with oxidative stress. TB and HIV/Aids are also diseases with chronic inflammation. The present study aims to evaluate the effects of NAC as a adjuvant therapy in the treatment of TB. This is a phase II randomized clinical trial in which the safety and tolerability of NAC as adjunctive therapy for TB treatment will be assessed. Fifty-six patients will be randomized into two groups. The first group will receive the standard tuberculosis treatment as recommended by the Brazilian Ministry of Health (RIPE); the second will receive in addition to this treatment 1200mg of NAC per day for two months. In this way, microscopy and culture conversion rate to mycobacteria at 8 weeks, levels of glutathione and biomarkers of immune activation and inflammation in case of TB with or without NAC will be monitored.

DETAILED DESCRIPTION:
TB and AIDS are also diseases that occur with a chronic inflammatory stimulus, with constant formation of excessive free radicals, leading to cellular and systemic oxidative stress. The effects of NAC in both populations are studied. A study demonstrated that HIV-positive individuals have low levels of glutathione in CD4+ T lymphocytes when compared to healthy controls, these levels being restored after in vivo supplementation with NAC, favoring the production of cytokines involved in Th1 response. They also observed that glutathione depletion in lymphocytes was correlated with increased levels of tumor necrosis factor and free radicals. Some authors suggested that the immune system's inability of HIV-positive individuals (or not) in containing Mycobaterium tuberculosis (Mtb) may be a consequence of low levels of glutathione in macrophages. The same occurred in a model of animals infected with Mtb, suggesting that oxidative stress was partly due to the poor antioxidant defense of the host. NAC supplementation decreases the bacterial load on the spleen and the severity of necrosis in the lung. The balance between oxidative and antioxidant substances plays a critical role in the induction of IL-12 production involved in the Th1 response and suggests that the use of NAC may be useful for better immune control of TB. Additional benefits of NAC in individuals with TB are related to the possible protective effect of hepatic to tuberculostatic drugs and to the direct antimicrobial effect demonstrated in vitro. Some authors suggest that the restoration of glutathione levels reversed the loss of innate immunity functions, pointing to a new mechanism of control of Mtb and a possible complement to antiretroviral treatment. This clinical trial will be undertaken in the Amazonas State (Western Brazilian Amazon), in Manaus, at Fundação de Medicina Tropical Dr. Heitor Vieira Dourado. It is a prospective, open-label, 2-arm, randomized clinical trial. Twenty-five patients will be enrolled in each treatment arm. A total number of 50 patients should be enrolled. Patients hospitalized in the ICU, in the wards or emergency room of the tertiary unit care will be invited to participate in this study. The assessment schedule will be done in days 1, 7, 14, 28, 42, 56, 120 and 180 (in addition, patient will be asked to come back to the health centre if symptoms occurs at any time). Sputum and blood collection and medical evaluation will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years;
* Acceptance of the HIV test;
* Forecast of hospital stay of more than twenty-four hours;
* Clinical and laboratory indication of RIPE;
* Conditions for puncture of venous access;

Exclusion Criteria:

* Brazilian indigenous people;
* People the refuse to perform HIV test;
* Pregnant women, nursing mothers or pregnant women,
* Extra pulmonary TB, without pulmonary involvement;
* Not be able to perform the collection of sputum or tracheal aspirate for microbiological confirmation;
* No MGIT® positive for Mtb;
* Resistance to Mtb, detected by professional sensitivity;
* Individuals under treatment for bronchospasm secondary to bronchial asthma, according to the decision of the assistant team or researcher of the study;
* Clinical suspicion of gastric or duodenal ulcer, as decided by the assistant team or study investigator; or evidence by upper digestive endoscopy;
* Alanine aminotransferase (ALT) greater than three times normal;
* Need to suspend the RIPE treatment, according to the decision of the assistant team or researcher of the study;
* Lack of adherence to the proposed treatment for more than seven consecutive days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-12-07 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with any biological intolerability or adverse event | 6 months
  This evaluation will be done by the physician along all the follow-up of the study

SECONDARY OUTCOMES:
Number of patients in the NAC treatment arm with shorter sputum smear conversion time and culture | Until week 8
  This outcome will be monitored by culture of solid (Löwenstein Jensen) and liquid (MGIT) sputum
Number of patients presenting tuberculostatic drug-related hepatotoxicity | 6 months
  This outcome will be monitored by hepatic transaminases and bilirubins levels
Dosage of inflammatory cytokines | 6 months
  This outcome will be evaluate immunological assays in the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo C dos Santos, MD, PhD, Principal Investigator — Fundação de Medicina Tropical Dr. Heitor Vieira Dourado; Bruno B Andrade, MD, PhD, Principal Investigator — Fundação Osvaldo Cruz Bahia
Locations (1):
- Fundação de Medicina Tropical Dr. Heitor Vieira Dourado, Manaus, Amazonas, Brazil

IPD SHARING:
Plan to Share IPD: No